CLINICAL TRIAL: NCT04679194
Title: Ph 1 Study of Escalating Single & Multiple Doses of Mana 312 (Multi Tumor-Associated Antigen T Cells) Administered to Adult Subjects With Acute Myeloid Leukemia or Myelodysplastic Syndrome After Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Study of Mana 312 (Multi Tumor-Associated Antigen T Cells) in Adults With AML/MDS After HSCT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Product manufacturing
Sponsor: Mana Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ManaTx-1001
Record Dates: First submitted 2020-12-14; First posted 2020-12-22 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: AML/MDS
Keywords: AML; MDS; Relapse; HSCT
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mana 312 (Experimental): Mana 312 is administered intravenously (IV) within 30 minutes in either an inpatient or outpatient setting; either a central or peripheral IV line may be used. Each cycle of administration of Mana 312 will be 28 days.
  Subjects not experiencing dose-limiting toxicity (DLT) following their initial dose may continue receiving their assigned Mana 312 dose every 28 days for an additional 2 doses
  Interventions: Biological: Mana 312

INTERVENTIONS:
Biological: Mana 312 — Mana 312 is a cellular product comprised of expanded T cells derived from allogeneic donor leukocytes that have been stimulated with monocyte derived dendritic cells pulsed with tumor-associated antigen (TAA) peptide mixes for 3 antigens: Wilms Tumor gene 1 (WT 1), the preferentially expressed antigen of melanoma (PRAME), and Survivin.
  Each Mana 312 product is specifically matched for an individual subject and will be manufactured from leukocytes from the same donor who provided stem cells to that subject for their current allogeneic hematopoietic stem cell transplantation (HSCT).

SUMMARY:
This is a Phase 1, open-label, non-randomized, single and multiple dose escalation study designed to evaluate the safety and preliminary efficacy of administering Mana 312 to subjects with AML/MDS after allogeneic HSCT.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, non-randomized, single and multiple dose escalation study designed to evaluate the safety and preliminary efficacy (prevention of, or treatment of relapse) of administering Mana 312 to subjects with AML/MDS after allogeneic HSCT. The study will evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of single and multiple doses of Mana 312. Each cycle of administration of Mana 312 will be 28 days.

In the Escalation Cohorts, subjects with low, intermediate, and adverse/high risk of relapse will be enrolled using a modified 3+3 design. Upon completion of Cycle 1, subjects not experiencing dose-limiting toxicity (DLT) may continue receiving their assigned Mana 312 dose every 28 days for an additional 2 doses unless the subject experiences progressive disease (PD), exhausts their supply of Mana 312, experiences intolerable side effects, is removed by the Investigator, withdraws consent, or the study is terminated. After Cohort 1 has been completed (i.e., a decision has been made to proceed to Cohort 2), enrollment will be limited to subjects with high-risk of relapse AML/MDS (see Inclusion Criterion #4b) until the RP2D is determined).

In the Expansion Cohort, only subjects with high risk of relapse AML/MDS will be enrolled using the RP2D of Mana 312. Subjects in the Expansion Cohort will receive Mana 312 at the time of relapse or at 1 year after HSCT, whichever is first. Subjects not experiencing dose-limiting toxicity (DLT) may continue receiving their assigned Mana 312 dose every 28 days for an additional 2 doses unless the subject experiences progressive disease (PD), exhausts their supply of Mana 312, experiences intolerable side effects, or the study is terminated.

ELIGIBILITY:
Select Inclusion Criteria:

1. Subject is ≥18 years of age on the day Informed Consent is signed and dated.
2. Subject must have received only one allogeneic HSCT from a related or unrelated donor prior to administration of Mana 312.
3. Subject has a donor who has agreed to donate leukocytes for manufacture of Mana 312 and who is the same donor who provided cells for the subject's current HSCT.
4. a. Prior to HSCT, for Escalation Cohort 1, subject has AML/MDS b. Prior to HSCT, for Escalation Cohorts after Cohort 1 and for the Expansion Cohort, a subject must have high risk of relapse AML/MDS
5. Mana 312 product is available

   The following Inclusion Criteria apply only during the Pre-Infusion Screening Phase, prior to the time of the planned first infusion of Mana 312.
6. Subject has Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3 or Karnofsky/Lansky score of ≥ 50.
7. Subjects in the Expansion Cohort must have a relapse of AML/MDS (MRD+ or morphologic relapse)
8. Subject has adequate organ function

Select Exclusion Criteria:

1. Subject has received antibody that affects T-cell number or function
2. Subject has received a donor lymphocyte infusion (DLI) for the current HSCT.
3. Evidence of GVHD ≥ Grade 2 in any organ system, or active bronchiolitis obliterans syndrome, sclerotic GVHD, or symptomatic serositis.
4. Subject has undergone major surgery (excluding minor procedures, eg, placement of vascular access, gastrointestinal/biliary stent, apheresis, or biopsy) < 21 days prior to the first planned infusion of Mana 312.
5. Subject has an active and clinically relevant infection
6. Subject has symptomatic or uncontrolled brain metastases, leptomeningeal disease, or spinal cord compression (radiation therapy to local site for disease control is allowed if ≥ 14 days prior to Screening and all AE from radiation therapy have resolved to ≤ Grade 1 prior to the planned first Mana 312 infusion).
7. Subject has any other medical condition not listed above or social condition that, in the opinion of the Investigator, might place the subject at increased risk, adversely affect compliance, or confound safety or other clinical study data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Escalation Cohorts: Identify the Maximum Tolerated Dose (MTD) of Mana 312 based on the safety and tolerability of single and multiple doses. | 6 months
  Maximum Tolerated Dose
Escalation Cohorts: Identify the Recommended Phase 2 Dose (RP2D) of Mana 312 based on the safety and tolerability of single and multiple doses. | 6 months
  Recommended Phase 2 Dose
Expansion Cohort: Assess preliminary antitumor efficacy of Mana 312 by CR. | 1 year
  CR Rate
Expansion Cohort: Assess preliminary antitumor efficacy of Mana 312 by PFS. | 1 year
  PFS Rate

SECONDARY OUTCOMES:
Escalation Cohorts: Assess preliminary evidence of Mana 312 antitumor efficacy by CR. | 1 year
  CR Rate
Escalation Cohorts: Assess preliminary evidence of Mana 312 antitumor efficacy by PFS. | 1 year
  PFS Rate
Expansion Cohort: Confirm safety of the RP2D by measurement of TEAEs. | 6 months
  Assess number of Treatment Related Adverse Events

OTHER OUTCOMES:
Characterize the pharmacokinetics (PK) by measurement of Mana 312 cell counts | 6 months
  Determine Mana 312 cell counts
Characterize the pharmacokinetics (PK) by measurement of antidrug antibodies (ADAs) | 6 months
  Measure presence or absence of antidrug antibodies to Mana 312
Characterize the anti-drug antibody (ADA) response to Mana 312. | 6 months
  Detect presence or absence of neutralizing antibodies to Mana 312
Determine Area Under the Curve (AUC) Pharmacokinetics of Mana 312 | 6 months
  AUC
Measure the Maximum Concentration Pharmacokinetics of Mana 312 | 6 months
  Cmax
Measure blast cell antigen expression pharmacodynamic markers of Mana 312 | 1 year
  Measure expression of three target antigens
Assess potential cytokine induction pharmacodynamic markers of Mana 312 | 1 year
  Assess potential cytokine induction as potential biomarker of pharmacodynamic activity
Measure cell expansion pharmacodynamic markers of Mana 312 | 1 year
  Measure cell expansion persistence of Mana 312 subclones
Measure immune subset pharmacodynamic markers of Mana 312. | 1 year
  Measure immune subset changes by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Lou Vaickus, MD, Principal Investigator — Mana Therapeutics Interim Chief Medical Officer
Locations (8):
- United States (8):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Northside Hospital - Atlanta, Atlanta, Georgia
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - Texas Transplant/St David's South Austin, Austin, Texas
  - Texas Transplant/Methodist Hospital, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No